CLINICAL TRIAL: NCT02269644
Title: A Phase 3, Double-blinded, Randomized, Comparator Trial of the Safety and Efficacy of a Single Dose of Dalbavancin to Twice Daily Linezolid for the Treatment of Community Acquired Bacterial Pneumonia
Brief Title: A P3 Comparator Trial in Community Acquired Bacterial Pneumonia
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Durata Therapeutics Inc., an affiliate of Allergan plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DUR001-305; 2014-002683-32 (EudraCT Number)
Record Dates: First submitted 2014-10-07; First posted 2014-10-21 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — dalbavancin; Linezolid; Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dalbavancin (Experimental): Dalbavancin randomized subjects will receive one dose of dalbavancin 1500 mg IV over 30 minutes on Day 1 plus azithromycin 500 mg IV on Day 1. Dalbavancin dose will be adjusted for subjects with significant renal insufficiency who are not receiving regular hemodialysis. All patients in the dalbavancin group will receive placebo linezolid infusions or tablets to maintain the blinding. Dalbavancin dose will be adjusted for subjects with significant renal insufficiency who are not receiving regular hemodialysis
  Interventions: Drug: Dalbavancin
- Linezolid (Active Comparator): Linezolid randomized subjects will receive linezolid 600 mg every 12 hours for a minimum of 10 days, and a maximum of 14 days. All patients will receive at least one IV dose of linezolid initially plus azithromycin 500 mg IV only on Day 1. Subjects then may then be switched to oral linezolid at the discretion of the investigator, if clinical improvement in the signs and symptoms of pneumonia is observed, to complete the 10-14 day course of therapy,. No dose adjustment is required for renal insufficiency.
  Interventions: Drug: Linezolid
- Linezold Placebo IV and Oral Capsules (Other): Dalbavancin randomized subjects after the 1st dose on Day 1 will receive placebo linezolid every 12 hours for a minimum of 10 days and a maximum of 14 days. Dalbavancin randomized subjects may be switched to oral linezolid placebo therapy to complete the 10-14 day course of therapy.
  Interventions: Drug: Linezolid Placebo
- Azithromycin (Other): Dalbavancin and linezolid randomized subjects on Day 1, 1st dose will also receive 500 mg of IV azithromycin
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Dalbavancin — dalbavancin 1500 mg IV over 30 minutes on Day 1
  Other Names: Dalvance
  Arms: Dalbavancin
Drug: Linezolid — linezolid 600 mg every 12 hours for a minimum of 10 days and a maximum of 14 days
  Other Names: Zyvox
  Arms: Linezolid
Drug: Linezolid Placebo — Dalbavancin randomized subjects after Day 1, 1st dose will receive linezolid placebo every 12 hours for a minimum of 10 days and a maximum of 14 days
  Arms: Linezold Placebo IV and Oral Capsules
Drug: Azithromycin — Dalbavancin and linezolid randomized subjects on Day 1, 1st dose receive 500 mg of IV azithromycin
  Arms: Azithromycin

SUMMARY:
This study will be a double-blind, randomized, multicenter trial to assess the safety and efficacy of a single 1500 mg IV dose of dalbavancin plus a single 500 mg IV dose of azithromycin in comparison to an approved antibiotic regimen of linezolid 600 mg every 12 hours for 10-14 days plus a single 500 mg IV dose of azithromycin for the treatment of Community Acquired Bacterial Pneumonia.

DETAILED DESCRIPTION:
This study will be a double-blind, randomized, multicenter trial to assess the safety and efficacy of a single 1500 mg IV dose of dalbavancin plus a single 500 mg IV dose of azithromycin in comparison to an approved antibiotic regimen of linezolid 600 mg every 12 hours for 10-14 days plus a single 500 mg IV dose of azithromycin for the treatment of CABP. Adult patients who meet all inclusion and none of the exclusion criteria will be randomized to one of the two treatment arms. Dosing will commence on Day 1, and all patients will receive a minimum of 10 days of therapy. Patients will be assessed on Day 1, Day 4-5, Day 7, Day 14 (End of Therapy, EOT), and Day 28 (Follow up).

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 to 85, inclusive
2. Has given written, informed consent
3. Has acute illness with onset within previous 7 days
4. Has at least 2 of the following symptoms:

   * Difficulty breathing or shortness of breath
   * Cough
   * Production of purulent sputum
   * Pleuritic chest pain
5. Has at least 2 vital sign abnormalities:

   * Fever (> 38°C or < 35°C)
   * Hypotension (systolic BP < 90 mm Hg)
   * Tachycardia (> 100 beats /min)
   * Tachypnea (> 24 breaths /min)
6. Has at least one other clinical or laboratory abnormalities:

   * Hypoxemia (room air SaO2 < 90% )
   * Clinical evidence of pulmonary consolidation
   * Elevated WBC count or neutropenia (> 12,000/mm3 or < 4,000/mm3)
7. Has new lobar or multi-lobar infiltrates on chest radiograph
8. Has CURB-65 risk category 1 to 4. Patients with CURB-65 risk category 1 will be limited to 20% of the total patient population

Exclusion Criteria:

1. Contra-indication to the administration of any of the study treatments, such as hypersensitivity to any of the glycopeptide agents, beta-lactam agents, linezolid or macrolide antibiotics, or current or recent (within 2 weeks) use of MAO inhibitors or serotonergic antidepressants (within 5 weeks for fluoxetine) (see Section 5.5.1)
2. Has received antibiotic therapy in the 4 days prior to screening, with the following exception: up to 25% of patients may have received a single dose of a short acting (half life < 8 hours) antibiotic
3. Has aspiration pneumonia
4. Has hospital acquired or ventilator associated pneumonia, or healthcare associated pneumonia, or 2 or more days in hospital in the previous 90 days
5. Has cystic fibrosis or known or suspected Pneumocystis pneumonia or known or suspected active tuberculosis
6. Females of child-bearing potential who are unable to take adequate contraceptive precautions, have a positive pregnancy result within 24 hours prior to study entry, are known to be pregnant, or are currently breastfeeding an infant
7. Has primary or metastatic lung cancer
8. Has known bronchial obstruction or a history of post-obstructive pneumonia
9. Requires admission to ICU at baseline
10. Has empyema requiring drainage
11. Infection due to an organism known prior to study entry to be resistant to either treatment regimen
12. Has known or suspected infection due solely to an atypical pathogen such as Mycoplasma sp., Chlamydia sp. or Legionella sp. or positive Legionella urinary antigen at baseline
13. Absolute neutrophil count < 500 cells/mm3
14. Known or suspected human immunodeficiency virus (HIV) infected patients with a CD4 cell count < 200 cells/mm3 or with a past or current acquired immunodeficiency syndrome (AIDS)-defining condition and unknown CD4 count
15. Patients with a recent bone marrow transplant (in post-transplant hospital stay)
16. Patients receiving oral steroids > 40 mg prednisolone per day (or equivalent) or receiving immunosuppressant drugs after organ transplantation
17. Patients with a rapidly fatal illness, who are not expected to survive for 3 months
18. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study
19. Has participated in another trial of an investigational pharmaceutical product in the 30 days prior to enrollment
20. Prior participation in this trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Treatment Response of CABP Symptoms | Change from Baseline to 72-120 hours after randomization
  Compare the efficacy of a single 1500 mg dose of intravenous dalbavancin plus azithromycin to the comparator regimen (linezolid plus azithromycin). Response will be based on resolution of symptoms; including chest pain, shortness of breath (difficulty breathing), frequency/severity of cough and amount of sputum production. Each of these symptoms will be assessed on a 4 point scale (absent, mild, moderate or severe). A patient will be defined as a clinical responder if there is at least a 1 point improvement in 2 or more of these symptoms at 72-120 hours after randomization compared to baseline.

SECONDARY OUTCOMES:
Efficacy of dalbavancin to the comparator regimen | Change from baseline to 72-120 hours after randomization, Day 14 and Day 28
  Test the efficacy of dalbavancin to the comparator regimen using alternative outcome measures including:1) improvement at Day 4-5 in at least two of the following symptoms with no worsening in any of these symptoms of CABP compared to baseline: chest pain, frequency or severity of cough, amount of productive sputum, and difficulty breathing and improvement in vital signs (i.e. temperature, heart rate, respiratory rate or blood pressure); 2) clinical outcome (using primary response criteria) at Day 14; 3) Investigator Assessment of Outcome at Day 14 and Day 28, with success defined as complete resolution of symptoms and signs attributable to CABP and did not receive non-trial antibacterial drugs for treatment of CABP.4) all-cause mortality at Day 28
Safety Analysis | Safety will be assessed at all time-points through Day 28
  To test the safety profile of dalbavancin 1500 mg versus comparator. Safety will be assessed by means of physical examination and vital signs, collection of adverse, events and clinical laboratory tests through out the study.

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — Durata Therapeutics Inc., an affiliate of Allergan plc
Locations (1):
- Mercury Street Medical Group, Butte, Montana, United States